CLINICAL TRIAL: NCT01289236
Title: An Exploratory, Randomized, Single Blinded, Placebo-Controlled, Dose-Ranging Study of the Safety and Efficacy of "MILNACIPRAN" in Subjects With Chronic Shoulder Pain
Brief Title: "MILNACIPRAN" in Subjects With Chronic Shoulder Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valera Bussell (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Valera Bussell, Sponsor Representative, Delray Research Associates
Organization: Delray Research Associates (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAV-MD-02
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Shoulder Pain
Keywords: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo BID (twice daily, approximately 12 hours apart)
  Interventions: Drug: Placebo
- milnacipran 200 mg (Active Comparator): 200mg- 1 100mg tablet BID (twice daily, approximately 12 hours apart)
  Interventions: Drug: Milnacipran
- milnacipran 100 mg (Active Comparator): 100mg- 1 50mg tablet BID (twice daily, approximately 12 hours apart)
  Interventions: Drug: milnacipran

INTERVENTIONS:
Drug: milnacipran — 1 tablet (50mg) BID (twice daily, approximately 12 hours apart) for 12 weeks after appropriate titration period
  Other Names: Savella
  Arms: milnacipran 100 mg
Drug: Milnacipran — 1 tablet (100mg) BID (twice daily, approximately 12 hours apart)for 12 weeks after appropriate titration period.
  Other Names: Savella
  Arms: milnacipran 200 mg
Drug: Placebo — 1 tablet (placebo) BID (twice daily, approximately 12 hours apart) for 12 weeks after appropriate titration period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of multiple doses of "Milnacipran" to a placebo dose in subjects with Chronic Shoulder Pain.

DETAILED DESCRIPTION:
16 weeks. It is planned that this study will be conducted at a single site and will enroll approximately 40 subjects over 2-4 months. At the end of the 12-week dosing period, the study drug will be discontinued and all subjects in the treatment groups and control group will be followed for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males, postmenopausal/ sterile females or females using reliable contraceptives who are >25 years of age.
2. Chronic shoulder pain in at least one shoulder for > 3 months (If both shoulders are painful, the investigator will choose the most painful shoulder for evaluation during the study) If both are equally painful, the investigator will choose the shoulder for evaluation.
3. History of shoulder or proximal arm pain due to bursitis, osteoarthritis of the shoulder, impingement or rotator cuff tear.
4. Subjects who give their written informed consent.
5. Subjects who at screening are not on chronic analgesic/anti-inflammatory medication and have a VAS pain score of > 40mm and < 90mm or subjects who are on chronic analgesic/anti-inflammatory medication at screening and have a VAS pain score of > 30mm and < 90mm, indicating a lack of adequate and sustained response to current therapy.
6. At baseline, after all analgesic/anti-inflammatory medication has been discontinued for 2 weeks (including withdrawal from acetaminophen rescue medication for 24 hours prior to screening) should have a VAS pain score of > 40mm and < 90mm.
7. Subjects who are willing to discontinue all NSAIDs or other analgesic medication taken for their shoulder pain with the exception of acetaminophen 500-1000mg (1-2 tablets) q.i.d., p.r.n. (maximum 8 tablets or 4 grams per day. Subjects must be willing to use only acetaminophen as a rescue pain medication for the shoulder pain. All analgesic medications must be stopped at least 2 weeks prior to the baseline visit and all acetaminophen must be discontinued at least 24 hours prior to the baseline visit. Subjects must be willing to abstain from any peri-articular injections for the shoulder during the course of the trial.
8. Subjects who have an x-ray at screening or MRI within 6 months prior to screening.

Exclusion Criteria:

1. Women of childbearing potential may not be entered if:

   Their pregnancy tests (urine) are positive They are nursing They do not use or agree to use an effective method of contraception until all follow-up procedures are complete. (Acceptable methods of contraception are oral, injectable, implanted contraceptive agent, abstinence or an intra-uterine device with a failure rate of < 1%
2. Participation in another experimental drug/device study within the past 30 days.
3. Acute infection of the study joint
4. History of adverse reaction or allergy to milnacipran or acetaminophen
5. Shoulder pain due to an injury for which litigation is planned or pending.
6. Any cervical spine disease that in the opinion of the investigator could confound assessments during the study.
7. Use of any oral corticosteroid during the past 30 days or peri-articular corticosteroid injection during the past 1 month.
8. Subjects with shoulder x-ray findings of fractures or avascular necrosis.
9. Subjects with any inter-current disease or condition that may interfere with the free use or evaluation of the affected shoulder for the duration of their participation in the study (severe congenital defects, weight bearing use of the shoulder due to crutches, walkers, canes etc.)
10. Subjects with history of alcohol or drug abuse within the past 5 years.
11. Subjects who have a compromised mental capacity or who may be unable to legally comprehend the details and nature of the study.
12. In the opinion of the investigator, a clinically significant abnormal lab results or history of disease that may place the subject at a health risk or compromise the study data or affect the subject's ability to complete the study.
13. Subjects who in the opinion of the investigator are unlikely to adhere to the study protocol or to complete the study as planned.
14. Subject has a chronic pain condition (chronic low back pain, chronic headache, fibromyalgia, chronic osteoarthritis, chronic rheumatoid arthritis etc.) that could confound the shoulder pain response to the study medication(in the opinion of the investigator)
15. Subject is using and is not willing to discontinue opioids, topical counterirritants (eg methylsalicylate or capsaicin) or the use of orthopedic devices for the study shoulder.
16. Significant liver impairment (defined as liver enzymes elevated more than three times the upper limit of normal) or significant renal impairment (defined as a serum creatinine level greater than twice the upper limit of normal.
17. Uncontrolled hypertension, history of stroke or transient ischemic attack within 6 months of enrollment, epilepsy, history of malignant neoplastic disease that is active (basal cell carcinoma of the skin is permitted), active infectious disease.
18. Subjects who have a history of uncontrolled Narrow Angle Glaucoma
19. Subjects who test positive for illegal or prohibited substances at Screening as demonstrated by a positive urine test or based on the Investigator's judgment.
20. Subjects who have active peptic ulcer disease, a history of inflammatory bowel disease or celiac sprue.
21. Subjects who have pulmonary dysfunction or severe chronic obstructive pulmonary disease that in the Investigator's opinion could interfere with study participation and completion.
22. Subjects who have unstable endocrine disease, including unstable diabetes or thyroid disease. Subjects with endocrine disorders that have been stable for the preceding 3 months will be permitted to enroll.
23. Male subjects with prostatic enlargement or other genitourinary disorders that put them at potentially significant risk for dysuria and/or urinary retention while taking agents with noradrenaline-reuptake inhibition properties (Entry permitted at Investigator's discretion)
24. Subjects who must participate in Physical Therapy during the course of their participation, unless stable in the opinion of the investigator.
25. Subjects with shoulder pain or other referred pain that does not originate from the shoulder.
26. Subjects who are taking SNRIs such as: Cymbalta
27. Subjects who are taking Lyrica or Neurontin
28. Subjects with cervical radiculopathy.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the reduction in the mean VAS for chronic shoulder pain | Week 12
  The primary efficacy endpoint will be the reduction in the mean VAS (Visual Analog Scale) for chronic shoulder pain at Week 12

SECONDARY OUTCOMES:
Improvement in the PGIC | Week 12
  Overall improvement in the PGIC (Patient Global Impression of Change) at Week 12
An improvement in the SPADI score | Week 12
  Improvement in the SPADI (Shoulder Pain and Disability Index) score at Week 12
Improvement in the SF-36 Health Questionnaire | Week 12
  Improvement in the SF-36 (Short Form-36) Health Questionnaire at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Saxe, MD,FACP, Principal Investigator — Delray Research Associates
Locations (1):
- Delray Research Associates, Delray Beach, Florida, United States